CLINICAL TRIAL: NCT00469469
Title: A Phase II Study of Bevacizumab in Patients With Nonresectable Cancer of the Adrenal Cortex.
Brief Title: Treatment Study Using Bevacizumab for Patients With Adrenocortical Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: unable to enroll subjects into the study
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Genentech, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMS 0510
Record Dates: First submitted 2007-05-02; First posted 2007-05-04 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2008-05

CONDITIONS: Adrenocortical Carcinoma
Keywords: Adrenal Cortex; ACC
MeSH Terms: conditions — Adrenocortical Carcinoma | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Bevacizumab

SUMMARY:
This is a Phase II study of intravenous Bevacizumab in patients with pathologically confirmed nonresectable primary adrenocortical cancer (ACC). Patients must have received no prior therapy. They will receive Bevacizumab as a single agent every 2 weeks intravenously until disease progression. This study will be open at multiple sites.

DETAILED DESCRIPTION:
Adrenocortical carcinoma(ACC)is a rare malignancy with an incidence of 1.5 to 2 per million per year in the United states. Surgery is the only therapeutic option that can prolong survival. Currently there are no therapies that have been proven to prolong survival for patients with nonsurgically resectable disease. ACC has been shown to be highly resistant to standard chemotherapy, therefore, it is important that we test agents with mechanisms of action. This is a single arm phase II study of Bevacizumab, an angiogenesis inhibitor, given as a single agent at 10 mg/kg IV every 2 weeks in patients with unresectable ACC. Bevicizumab will be used as first line therapy. The study will test if Bevacizumab will be able to prolong the time to progression. If a delay in time to progression of 4 months or greater is seen, this will be considered clinically meaningful and further studies will be considered. This study will be conducted at multiple institutions (see below).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide written informed consent
* Subjects must be 18 years of age or older
* Subjects must have histologically confirmed ACC by the Department of Pathology at Dartmouth-Hitchcock Medical Center
* Subjects must have inoperable disease
* This is a first and/or second line study. Patients must have completed only one or fewer regimes of systemic therapy. They may have received one prior systemic therapy either: a) mitotane, or b)chemotherapy, or c) experimental therapy, or d) concurrent chemotherapy and mitotane, or e) no prior systemic therapy
* Subjects must have a life expectancy of three or more months
* If subjects have received some form of systemic therapy (e.g. chemotherapy or mitotane), they should have completed that systemic therapy at least 28 days before beginning Bevacizumab
* All subjects of child-bearing potential(men and women) must agree to the use of effective means of contraception

Exclusion Criteria:

* Other co-existing malignancies or malignancies diagnosed within the last 5 years wtih the exception of basal cell carcinoma or cervical cancer in situ
* Any unresolved chronic toxicity greater than CTC grade 2 from previous anticancer therapy (except alopecia)
* absolute neutrophil counts less than 1.5 x l,000,000,000/liter, or platelets less than 20.0 x 1,000,000,000/liter
* As judged by the investigator, any evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory,cardiac, hepatic, or renal disease)
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the trial
* Prior therapy with two or more systemic therapy regimes. In other words if a patient is seeking third line therapy or later than third line therapy he is ineligible for this study
* Current, recent(within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech- sponsored Bevacizumab cancer study
* Prior use of Bevacizumab or any other anti-VEGF therapies
* Known hypersensitivity to Bevacizumab
* Inadequately controlled hypertension (defined as systolic blood pressure of >150 mm Hg and/or diastolic blood pressure >100 mm Hg on anti- hypertensive medications
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* Unstable angina
* New York Heart Association (NYHA)Grade II or greater congestive heart failure
* History of myocardial infarction within 6 months
* History of stroke or transient ischemic attack at any time prior to study enrollment
* Clinically significant peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Presence of central nervous system or brain metastases
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during the course of the study
* Core biopsies or other minor surgical procedures, excluding placement of a vascular access device, within 7 days prior to Day 0
* Pregnant (positive pregnancy test) or lactating
* Women who are fertile and not willing to practice abstinence or an adequate form of contraception (i.e. use or oral contraceptives, intrauterine devices or barrier protection)
* Urine protein: creatinine ratio > 1.0 at screening -History of abdominal fistula, gastrointestinal perforation, or intr- abdominal abcess within 6 months prior to Day 0
* Serious, non-healing wound, ulcer, or bone fracture
* Lung lesions of any etiology(malignant or nonmalignant) in close proximity to a major vessel
* Cavitary lung lesions (to prevent episodes of potentially life-threatening hemoptysis)
* History of hemoptysis (defined as bright red blood of 1/2 teaspoon or more)
* Inability to comply with study and/or follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-05; Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
To measure time to progression | From date of first dose of Bevacizumab until progression.

SECONDARY OUTCOMES:
To Measure objective response rate by RECIST | At the end of treatment, RECIST criteria will be used to determine the patient's best overall response.
To determine an adverse event profile | Measured from date of first treatment until 30 days post treatment.
To measure survival in all treated patients. | Survival is measured from the date of first treatment to date of death form any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Samnotra, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States